CLINICAL TRIAL: NCT06980870
Title: Effect of Pre-medication With Anti-inflammatory Drugs(Ibuprofen and Dexamethasone)on Post-Endodontic Pain With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Pre-medication With Anti-inflammatory Drugs(Ibuprofen and Dexamethasone)on Post-Endodontic Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Qurat-ul-ain Abbasi, Post-Graduate Resident Operative Dentistry & Endodontic, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ibuprofen versus Dexamethasone
Record Dates: First submitted 2025-02-15; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-02

CONDITIONS: Post-endodontic Pain; Ibuprofen; Dexamethasone
Keywords: post-endodontic pain; ibuprofen; dexamethasone
MeSH Terms: interventions — Anti-Inflammatory Agents; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pain with ibuprofen (Active Comparator): Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain
  Interventions: Drug: Anti-inflammatory drug (ibuprofen)
- Pain with dexamethasone (Active Comparator): Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain
  Interventions: Drug: Anti-inflammatory drug (dexamethsaone)

INTERVENTIONS:
Drug: Anti-inflammatory drug (ibuprofen) — Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain
  Arms: Pain with ibuprofen
Drug: Anti-inflammatory drug (dexamethsaone) — Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain
  Arms: Pain with dexamethasone

SUMMARY:
Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain with symptomatic irreversible pulpitis

DETAILED DESCRIPTION:
Study will be conducted after the approval of Institutional Ethics Review Committee, AFID (ANX "A").

A total of 130 entitled patients reporting to Operative Dentistry Department, Armed Forces Institute of Dentistry will be invited for participation in this study. The procedure will be explained to the patients and their parents in Urdu language and a written informed consent will be taken (ANX "B") They will be screened for inclusion by taking history, performing relevant clinical examination and necessary tests along with peri-apical radiographs. Patients fulfilling the inclusion criteria will be divided into two groups using consecutive non random sampling.

Group 1: Patients treated with premedication of Non steroidal anti inflammatory drug (Ibuprofen) Group 2: Patients treated with premedication of Steroidal anti inflammatory drug (Dexamethsone)

Both groups will receive medication 15 mins before intiating root canal treatment. Root canal treatment will then be initiated under local anesthesia and rubber dam isolation. Working length will be taken 1mm from radiographic apex with apex locator and will be confirmed with radiograph. The root canals will be instrumented with ProTaper Next system under copious irrigation with 5.25% sodium hypochlorite (NaOCl). Patency will be confirmed with a #10 K file between each instrument change. The root canals will be flushed with 5 mL of 17% EDTA solution. To control the microbiological impact on post-operative pain calcium hydroxide will be used as an intra-canal medicament and likewise 5.25% sodium hypochlorite as an irrigant in both groups. Following instrumentation and calcium hydroxide placement in the canal using lentulo spirals, the cavity will be temporarily sealed with cavit.

At the end of every appointment, patient will be given a visual analogue scale. The patient will be advised to mark the line corresponding with the intensity of his pain at 24, 48 and 72 hours after the first visit. The patient will be recalled after one week for obturation and final full coverage restoration. Analgesics will be prescribed in case of severe intolerable pain.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent teeth with acutely inflamed pulp without swelling or draining sinus.
2. Patients of either gender aged between 18-50 years old.
3. Systemically healthy patients.
4. Patients who agree to attend for recall appointments and provide a written consent.

Exclusion Criteria:

1. Patients on preoperative analgesics and antibiotics.
2. Teeth with calcified canals and previously treated teeth.
3. Pregnant and lactating mothers.
4. Patients who are immunocompromised, anxious and mentally handicapped.
5. Patients who are allergic to any of the test medications.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
effect of pre-medication(ibuprofen and dexamethasone ) on post-endodontic pain | 24 hours
  Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain on visual analogue scale
effect of pre-medication(ibuprofen and dexamethasone ) on post-endodontic pain | 48 hours
  Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain on visual analogue scale
effect of pre-medication(ibuprofen and dexamethasone ) on post-endodontic pain | 72 hours
  Effect of pre-medication with anti-inflammatory drugs(ibuprofen and dexamethasone)on Post-Endodontic pain on visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Quratulain Abbasi, BDS, Principal Investigator — AFID
Locations (1):
- Armed Forces Institute Of Dentistry, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided